CLINICAL TRIAL: NCT06178172
Title: Implementation of a Remote Home Monitoring Program for Patients With a Mild Acute Pancreatitis - A Single Center Feasibility Study
Brief Title: Remote Home Monitoring in Mild Acute Pancreatitis
Acronym: INTERACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rijnstate Hospital (Other)
Collaborators: University of Twente (Other); Philips Research Eindhoven (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL84869.100.23
Record Dates: First submitted 2023-11-30; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Pancreatitis, Acute; Remote Home Monitoring; Early Discharge
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early discharge with remote home monitoring. (Experimental): After at least 48 hours of hospital admission, patients are discharged early with the use of remote home monitoring. At home, patients receive guidance for the management of pain, nutrition and pancreatitis-related complaints by a daily phone call from a nurse from the Virtual Monitoring Centre (VMC). The pancreatitis-related complaints, intake of fluids and food, pain and the use of analgesics are assessed using short questionnaires in a smartphone app. Core temperature is monitored using an ear thermometer and a wearable sensor measures heart rate, respiratory rate, posture and movement every 5 minutes. Remote home monitoring will continue for at least 4 days.
  Interventions: Other: Remote home monitoring

INTERVENTIONS:
Other: Remote home monitoring — After at least 48 hours of hospital admission, patients are discharged early with the use of remote home monitoring. At home, patients receive guidance for the management of pain, nutrition and pancreatitis-related complaints by a daily phone call from a nurse from the Virtual Monitoring Centre (VMC). The pancreatitis-related complaints, intake of fluids and food, pain and the use of analgesics are assessed using short questionnaires in a smartphone app. Core temperature is monitored using an ear thermometer and a wearable sensor measures heart rate, respiratory rate, posture and movement every 5 minutes. Remote home monitoring will continue for at least 4 days.

SUMMARY:
Acute pancreatitis is an inflammation of the pancreas which causes abdominal pain and is the most common gastro-intestinal reason for acute hospitalization in Western countries. Because care for patients with a mild acute pancreatitis is mostly supportive, providing this care in the home environment may be feasible with the use of remote monitoring. This might reduce the demand for hospital beds and allow patients to benefit from recovering in their home environment. Therefore, the objective of this single center study is to assess the feasibility of a novel care program in which patients with a predicted mild course of acute pancreatitis are discharged early with remote home monitoring.

Patients, with a predicted mild course of acute pancreatitis. Patients with prior acute pancreatitis within 3 months or a chronic pancreatitis are excluded from participation. Patients should be ≥18 years of age. The goal is to include a total of 70 patients. After at least 48 hours of hospital admission, patients are discharged early with the use of remote home monitoring. At home, patients receive guidance for the management of pain, nutrition and pancreatitis-related complaints by a daily phone call from a nurse from the Virtual Monitoring Centre (VMC). The pancreatitis-related complaints, intake of fluids and food, pain and the use of analgesics are assessed using short questionnaires in a smartphone app. Core temperature is monitored using an ear thermometer and a wearable sensor measures heart rate, respiratory rate, posture and movement every 5 minutes. Remote home monitoring will continue for at least 4 days.

The main study objective is to assess the feasibility of the novel care program. Feasibility is determined by, patient satisfaction and actual use of the novel care program. The secondary study objective is to describe clinical outcomes of patients in the novel care program.

ELIGIBILITY:
Inclusion Criteria:

* Acute pancreatitis according to the revised Atlanta criteria for pancreatitis(23). Which is at least 2 of the following 3 criteria:

  * Abdominal pain consistent with acute pancreatitis
  * Serum lipase ≥ 3x upper limit normal (> 159 U/l)
  * Typical pancreatic abnormalities on imaging (ultrasound, CT or MRI)
* First episode of acute pancreatitis or a prior pancreatitis more than 3 months ago
* Age ≥18 years, both men and women
* Able and willing to provide written informed consent in Dutch
* In possession of a working (smart)phone on which patient can be reached for the duration of participation (30 days)
* ≤1 SIRS criteria

  * Temperature < 36◦C or > 38◦C
  * Heart rate >90/min
  * Respiratory rate >20/min
  * Leucocytes < 4x/109/L or > 12x109/L
* Serum CRP ≤ 150 mg/l on day of discharge and with a decreasing trend in days before
* Pain score (NRS) ≤6 with or without the use of pain medication
* Adequate intake of oral food and fluids (= ≥2 small meals and ≥1L fluids per day)
* Stable serum creatinine and Ringer's lactate infusion reduced to ≤1L/24 hours
* Independent in performing general daily life activities

Exclusion Criteria:

* Chronic pancreatitis according to M-ANNHEIM criteria(24).
* Acute cholangitis
* Endoscopic retrograde cholangiopancreatography within the first 24 hours of admission
* MEWS (Modified Early Warning Score) ≥6 or in need of ICU admission
* Living in an institution (e.g. psychiatric ward or nursing home), or the absence of a household member capable of alerting the hospital in case of an emergency Known sensitivity to medical adhesives
* Known pregnancy
* Have one or more of the following comorbidities:

  * Heart failure (NYHA class III or IV)
  * COPD (Gold III-IV)
  * Kidney disease (>G3b) and/or kidney replacement therapy
  * Currently undergoing oncological treatment
  * Use of immunosuppressants
  * Dysregulated or poorly controlled insulin dependent diabetes
  * Morbid obesity (BMI>35 kg/m2)
  * Implantable Cardioverter Defibrillator (ICD) or Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-10-02 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with overall care, based on satisfaction questionnaire | Within 30 days of hospital admission
  Overall care from GE-ward admittance until discontinuation of remote home monitoring.
Patient satisfaction with smartphone app (Luscii), based on satisfaction questionnaire | Within 30 days of hospital admission
Patient satisfaction with wearable sensor (Healthdot), based on satisfaction questionnaire | Within 30 days of hospital admission
Patient intent to participate in the care program again | Within 30 days of hospital admission
  Based on satisfaction questionnaire
Proportion of patients willing and able to participate | Within 30 days of hospital admission
Time between discharge decision and actual hospital discharge in days | Within 30 days of hospital admission
Duration of remote home monitoring in days | Within 30 days of hospital admission
Number of contacts between patients and healthcare professionals | Within 30 days of hospital admission
Number of additional laboratory tests (during home monitoring) | Within 30 days of hospital admission
Smartphone app functionality, determined by generated notifications, time between notification and contact with VMC-nurse and questionnaire compliance | Within 30 days of hospital admission
Wearable sensor functionality, determined by the amount of missing data and accidental detachments | Within 30 days of hospital admission

SECONDARY OUTCOMES:
Use of analgesics and anti-emetics, described as the number of days used | Within 30 days of hospital admission
Pain scores, based on NRS (0-10) | Within 30 days of hospital admission
Intake of food and fluids, described as number of meals and liters of fluid intake | Within 30 days of hospital admission
Activity levels, as measured by the wearable sensor (0-10) | Within 30 days of hospital admission
Time between GE ward admission and discharge decision in days | Within 30 days of hospital admission
Hospital readmissions | Within 30 days of hospital admission
Emergency department (ED) revisits | Within 30 days of hospital admission
  An ED revisit followed by a hospital readmission will be documented as a hospital readmission
Pancreatitis-related complications | Within 30 days of hospital admission
  Pseudocysts, necrosis, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Rijnstate Hospital, Arnhem

IPD SHARING:
Plan to Share IPD: Undecided
Data available upon reasonable request.